CLINICAL TRIAL: NCT06443853
Title: A Novel Approach to Digital Dental Plaque Scoring
Brief Title: Creating Digital Dental Plaque Scoring
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: Digital Scoring
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Dental Plaque
Keywords: dental plaque; dental plaque scoring; dental plaque imaging
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Clinical scoring: The Turesky Modified Quigley Hein Plaque Index of anterior teeth of the volunteers' was recorded using clinical visual examination after dental plaque staining.
  Interventions: Diagnostic Test: Dental plaque scoring and dental plaque coated tooth surface measuring
- Digital Camera: Intraoral photographs of the volunteers were taken by using a digital camera (Canon EOS 700D; 100 mm macrolens, Canon Inc., Tokyo, Japan).
  All taken photographs were transferred to the Image J V1.53 (National Institute for Health, Bethesda, USA) program. The plaque-covered area and the total surface area of the teeth were marked in the manual mode of the program.
  Interventions: Diagnostic Test: Dental plaque scoring and dental plaque coated tooth surface measuring
- Intraoral Scanner: 3D images of the volunteers were recorded by an intraoral scanner (iTero Element Flex, Align Technologies, San Jose, California, USA).
  All taken images were transferred to the Image J V1.53 (National Institute for Health, Bethesda, USA) program. The plaque-covered area and the total surface area of the teeth were marked in the manual mode of the program.
  Interventions: Diagnostic Test: Dental plaque scoring and dental plaque coated tooth surface measuring

INTERVENTIONS:
Diagnostic Test: Dental plaque scoring and dental plaque coated tooth surface measuring — The Turesky Modified Quigley Hein Plaque Index of anterior teeth of the volunteers' was recorded using clinical visual examination.
  Intraoral photographs of the volunteers were taken by using a digital camera and 3D images were recorded by an intraoral scanner. The plaque-covered area and the total surface area of the teeth were marked in the manual mode of the Image J program and the areas were measured in square pixels. The correlation between clinical visual scoring, dental plaque areas on images were compared.

SUMMARY:
It is aimed to compare dental plaque area measured on images obtained in the clinic by using dental photography and intraoral scanner and to evaluate the correlation of this area with clinical plaque scores.

Clinical dental plaque scoring was measured according to the "Turesky Modified Quigley Hein Plaque Index" after applying a plaque staining agent (Tri Plaque ID Gel, GC Corp., Tokyo, Japan) to evaluate the oral hygiene of 20 patients who applied to the university clinic. Following clinical scoring, intraoral photographs of the patients were taken using dental photography equipment of the same standards (EOS700D, Canon; 100mm lens, Canon; twin flash, Yong Nuo) and scan images were taken with an intraoral scanner (iTero Element Flex, Align Tech., USA). In the data obtained, dental plaque area on the buccal surface of 66 lower and upper jaw anterior teeth were measured with Image J (National Institute for Health, Bethesda, USA) software, and the ratio of dental plaque area to the visible surface area of the tooth was measured.

DETAILED DESCRIPTION:
The (h1) hypothesis of this study was that dental plaque scores measured through digital camera and intraoral scanner images can replace clinical visual scoring. This study aimed to compare dental plaque areas measured on images taken by digital camera and intraoral scanner and to evaluate these areas with clinical plaque scores with the help of a software program and provide a novel plaque index to score dental plaque on the taken intraoral images.

Study Design The tooth arches of the volunteers were stained with a plaque-disclosing solution (Tri Plaque ID Gel, GC Corporation, Tokyo, Japan). The Turesky Modified Quigley Hein Plaque Index (TMQHPI) of anterior teeth of the volunteers' was recorded using clinical visual examination.

Intraoral photographs of the volunteers were taken by using a digital camera (Canon EOS 700D; 100 mm macrolens, Canon Inc., Tokyo, Japan), and 3D images were recorded by an intraoral scanner (iTero Element Flex, Align Technologies, San Jose, California, USA). Photograph and intraoral scanner images were overlapped and pixel-synchronized using the Keynote program.

After synchronization, all taken images were transferred to the Image J V1.53 (National Institute for Health, Bethesda, USA) program. The plaque-covered area and the total surface area of the teeth were marked in the manual mode of the program and the areas were measured in square pixels. Measurements were made on a total of 66 teeth, which can be easily seen on the images. Intraoral scanner plaque area/ tooth surface area ratio and intraoral photograph plaque area/ tooth surface area ratio were calculated and recorded for each tooth.

ELIGIBILITY:
Inclusion Criteria:

* Patients without orthodontic brackets, fixed or implant restorations and without severe tooth crowding were included in the study.

Exclusion Criteria:

* Among the patients with orthodontic brackets, severe tooth crowding that could not be visually verified on images, fixed or implant restorations were excluded in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study included 20 patients between the age of 18 to 45. Among the patients with orthodontic brackets, severe tooth crowding that could not be visually verified on images, fixed or implant restorations were excluded in the study. Measurements were made on a total of 66 teeth, which can be easily seen on the images.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Correlation between Turesky Modified Quigley Hein Plaque Scores and dental plaque coated surface areas on the images taken by digital camera and intraoral scanner | 1 month
  The Turesky Modified Quigley Hein Plaque Index (TMQHPI) of anterior teeth of the volunteers' was recorded using clinical visual examination.Intraoral photographs of the volunteers were taken by using a digital camera and 3D images were recorded by an intraoral scanner.The plaque-covered area and the total surface area of the teeth were marked in the manual mode of the Image J program and the areas were measured.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Tagtekin, Professor, Study Director — Marmara University
Locations (1):
- Marmara University, Department of Restorative Dentistry, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided